CLINICAL TRIAL: NCT06252402
Title: A Pilot Study to Evaluate the Feasibility and Safety of Cytomegalovirus-Specific, Anti-HIV Chimeric Antigen Receptor (CMV-HIV CAR) T Cells in People Living With HIV
Brief Title: CMV-specific HIV-CAR T Cells as Immunotherapy for HIV/AIDS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22508
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: HIV-1
Keywords: HIV-1, PLWH (Healthy People Living with HIV-1) autologus; CMV-specific T cells, anti-retroviral therapy (ART), Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level -1 (Experimental): EGFR+ T Cell Dose (Day 0) 5 x 10^6 cells
  Interventions: Biological: CMV/HIV-CAR T Cells
- Dose Level +1 (Experimental): EGFR+ T Cell Dose (Day 0) 25 x 10^6 cells
  Interventions: Biological: CMV/HIV-CAR T Cells
- Dose Level +2 (Experimental): EGFR+ T Cell Dose (Day 0) 50 x 10^6 cells
  Interventions: Biological: CMV/HIV-CAR T Cells

INTERVENTIONS:
Biological: CMV/HIV-CAR T Cells — Eligible participants will temporarily interrupt their ART regimen for 4 days prior to leukapheresis to prevent residual cell drug levels that could inhibit lentiviral transduction of the T cells during CAR T cewll manufacturing. Participants will resume their ART regimen immediately after leukapheresis. Once the final cell product is released, participants will receive a single intravenous (IV)infusion of autologous CMV/HIV-CAT T cells (defined as Day 0). Up to three doses of CMV/HIV-CAR T cewlls may be explored.

SUMMARY:
Human immunodeficiency virus type 1 (HIV-1) causes a persistent infection that ultimately leads to acquired immunodeficiency syndrome (AIDS). Treatment of HIV-1 infection with combination anti-retroviral therapy (ART) suppresses HIV-1 replication to undetectable viral levels and saves lives. Nevertheless, ART cannot eradicate latent cellular reservoirs of the virus, and HIV-1 infection remains a life-long battle. Adoptive cellular immunotherapy using chimeric antigen receptor (CAR) engineered T cells directed against HIV-1 envelope subunit protein gp120 (HIVCAR T cells) may provide a safe and effective way to eliminate HIV-infected cells.

However, the number of HIV-infected cells is low in participants under ART, and CAR T cells disappear if they are not stimulated by their target antigens. Interestingly, about 95% of HIV-1-infected individuals are CMV-seropositive and CMV-specific T cells have been shown to persist. To overcome the CAR T cells low persistence issue, we propose to make HIV-CAR T cells using autologous cytomegalovirus (CMV)-specific T cells, which can be stimulated by endogenous CMV in vivo. The overall hypothesis of this first-in-human Phase 1, open-label, single-arm study is that endogenous immune signals to CMV-specific T cells can maintain the presence of autologous bispecific CMV/HIV-CAR T cells in healthy people living with HIV-1 (PLWH), and achieve long-term remission in the presence of ART.

DETAILED DESCRIPTION:
Human immunodeficiency virus type 1 (HIV-1) causes a persistent infection that ultimately leads to acquired immunodeficiency syndrome (AIDS). Treatment of HIV-1 infection with combination anti-retroviral therapy (ART) suppresses HIV-1 replication to undetectable viral levels and saves lives. Nevertheless, ART cannot eradicate latent cellular reservoirs of the virus, and HIV-1 infection remains a life-long battle. Adoptive cellular immunotherapy using chimeric antigen receptor (CAR) engineered T cells directed against HIV-1 envelope subunit protein gp120 (HIV-CAR T cells) may provide a safe and effective way to eliminate HIV-infected cells. However, HIV-infected cells in participants under ART, and CAR T cells disappear if they are not stimulated by their target antigens. Interestingly, about 95% of individuals with HIV-1 are CMV-seropositive and CMV-specific T cells have been shown to persist at high frequency due to CMV antigen stimulation. To overcome the CAR T cells low persistence issue, we propose to make HIV-CAR T cells using autologous cytomegalovirus (CMV)-specific T cells, which can be stimulated by endogenous CMV in vivo. The overall hypothesis of this first-in-human, open-label, single-arm, pilot study is that endogenous immune signals to CMV-specific T cells can maintain the presence of autologous bispecific CMV/HIV-CAR T cells in healthy people living with HIV-1 (PLWH). Based on the results of this safety study, CMV vaccine and analytic treatment interruption will be evaluated with the CMV/HIV-CAR T cell investigational product in a subsequent protocol.

The trial is a first-in-human, pilot study to evaluate the feasibility and safety and determine the maximum tolerated dose (MTD)/recommended Phase II dose (RP2D) of CMV/HIV-CAR T cells in PLWH. Eligible participants will temporarily interrupt their ART regimen for 4 days prior to leukapheresis to prevent residual cell drug levels that could inhibit lentiviral transduction of the T cells during CAR T cell manufacturing. Participants will resume their ART regimen immediately after leukapheresis. If the manufacturing is not successful, a second apheresis may be scheduled no sooner than 3 weeks later with temporary interruption of ART regimen for 4 days prior to leukapheresis. Participants will resume their ART regimen immediately after leukapheresis. Once the final cell product is released, participants will receive a single intravenous (IV) infusion of autologous CMV/HIV-CAR T cells (defined as Day 0). Up to three doses of CMV/HIV-CAR T cells may be explored.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age at the time of screening;
* Karnofsky Performance Status (KPS) ≥ 70;
* Documented HIV-1 infection anytime prior to study entry.;
* On stable ART with undetectable HIV-1 RNA (i.e < 20 copies /mL) for at least 48 weeks prior to screening (2 plasma HIV-1 RNA blips 25-200 copies/mL are allowable);
* CD4+ cell count ≥ 450 cells/μL;
* Adequate organ function;
* Willingness to interrupt ART regimen for 4 days prior to leukapheresis;
* Not pregnant or breastfeeding.

Exclusion Criteria:

* Concurrent illness or comorbid condition;
* History of resistance to two or more classes of antiretroviral drugs;
* History of prior receipt of an experimental HIV-1, immunotherapeutic agent, or gene therapy product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | Up to 28 days after the infusion
  Toxicity will be graded per CTCAE v5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Criteria on CRS/Neurotoxicity: DLT.
Toxicity profile | Up to 28 days after the infusion
  Toxicity will be graded per CTCAE v5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Criteria on CRS/Neurotoxicity: all other toxicities to define the toxicity profile.

SECONDARY OUTCOMES:
CD4+ T cell count and HIV RNA levels | Up to 28 days after the infusion
  CD4+ T cell count and HIV RNA levels in the peripheral blood;
EGFR+ CD3+ T cells | Up to 28 days after the infusion
  Number, percentage and persistence of EGFR+ CD3+ T cells in the peripheral blood and EGFR- CD3+ T cells in peripheral blood
Cytokine levels | Up to 28 days after the infusion
  Cytokine levels in the peripheral blood post CAR T cell infusion.
Number of CMV/HIV-CAR T cells | Up to 28 days after the infusion
  Number of CMV/HIV-CAR T cells: measured by qPCR in peripheral blood); and Using two in-depth interviews (1) shortly following screening (within 2 weeks), and 2) within 1 month of initiating Step 4, we will assess perceptions of the CMV/HIV-CAR T cell intervention and overall trial experiences in participants

CONTACTS AND LOCATIONS:
Overall Officials: John H. Baird, MD, Principal Investigator — City of Hope Medical Center; David (Davey) Smith, MD, Principal Investigator — UCSD, San Diego Center for AIDS Research
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - UCSD, Division of Infectious Diseases and Global Public Health, San Diego, California

IPD SHARING:
Plan to Share IPD: No